CLINICAL TRIAL: NCT03919188
Title: Comparison of Air vs. Cutaneous Control Mode for Preterm Infants ≤ 32 WG Raised in Closed Incubators: Impact on Body Growth and Morbidity
Brief Title: Air vs. Cutaneous Control Mode for Preterm Infants ≤ 32 WG in Incubators: Impact on Body Growth and Morbidity
Acronym: ThermoKPreterm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Caen (Other); University Hospital, Lille (Other); Centre Hospitalier Arras (Other); Centre Hospitalier de Montreuil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0056
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Preterm Infant; Body Temperature
Keywords: preterm neonates; incubator management; body temperature; relative air humidity; thermoneutrality
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- air temperature control (ATC) (Active Comparator): Incubator control using air temperature control (ATC) method
  Interventions: Procedure: air temperature control (ATC)
- skin servocontrol (SSC) (Active Comparator): Incubator control using skin servocontrol method
  Interventions: Procedure: skin servocontrol (SSC)

INTERVENTIONS:
Procedure: air temperature control (ATC) — Currently there are no guidelines for setting incubator parameters. The Cochrane database point out for further research (Sinclair, 2002). The investigators aim at evaluating 3 different incubator settings for the INOTHERM incubator (Mediprema, France): second parameter : air temperature control (ATC)
  Arms: air temperature control (ATC)
Procedure: skin servocontrol (SSC) — Currently there are no guidelines for setting incubator parameters. The Cochrane database point out for further research (Sinclair, 2002). The investigators aim at evaluating 3 different incubator settings for the INOTHERM incubator (Mediprema, France): Third parameter : skin servocontrol (SSC).
  Arms: skin servocontrol (SSC)

SUMMARY:
Previous studies have shown that mortality and morbidity in preterm neonates are correlated with the fall in body temperature on admission. Hypothermia can be decreased by reducing body heat losses to the environment. The investigator research hypothesis is that a new calculation of the air temperature in the incubator would promote the newborn infant weight growth from the period between birth and day 10 of life compared to cutaneous mode. The secondary hypotheses assumes a decrease in the side effects usually observed in both morbidity and mortality.

A software is used to calculate the body heat loss (BHL) of each individual preterm infant, and to propose a specific air temperature setting inside the incubator to reduce BHL to zero. This software has been validated in a previous pilot study (Degorre et al. 2015). This study aims to compare the energy costs of providing incubated preterm infants born between 25 and 32 weeks of gestation with homeothermia using either specific individualized air temperature control (ATC) or skin servocontrol (SSC).

ELIGIBILITY:
Inclusion Criteria:

* preterm infant born between 25+0 and 32+0 weeks of gestation
* preterm infant included in the study before 24 +/- 12 hours of life
* preterm infant nursed in a closed incubator
* written informed consent from his parents

Exclusion Criteria:

* newborn infant with polymalformative syndrome
* life threatening events or serious heart disease

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | until day 10 of life
  Change in body weight between birth and day 10 of life

SECONDARY OUTCOMES:
Comfort of the preterm infant | until day 10 of life
  Comfort of the preterm infant will be estimated by using the newborn infant physical examination (NIPE)
thermal stress occurence | until day 10 of life
  Thermal stress are hyperthermia rate, hypothermia rate, mean time in thermal comfort= thermal challenge
humidity challenge using TEWL | until day 10 of life
  TEWL = transepidermal water loss. It is a daily skin monitoring of hydric loss
neonatal morbidity occurence | until age corresponding to 40 weeks of amenorrhea
  neonatal morbidities are infectious rate, necrotizing enterocolitis (NEC), Intraventricular hemorrhage (IVH), Bronchopulmonary dysplasia (BPD) and death
length of hospitalization stay | until age corresponding to 40 weeks of amenorrhea or end of hospitalization
  length of hospitalization stay (number of days of hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Cénéric, Dr, Principal Investigator — CHU CAEN; Kévin Leduc, Dr, Principal Investigator — CHRU LILLE; Sophie Galène, MD, Principal Investigator — CHU Rouen; Guillaume ESCOURROU, MD, Principal Investigator — CHI André Grégoire - Montreuil; Julien Ghesquière, MD, Principal Investigator — CH Arras
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No